CLINICAL TRIAL: NCT01757639
Title: A Phase 1 Study of Ipilimumab in Relapsed and Refractory High Risk Myelodysplastic Syndrome and Acute Myeloid Leukemia With Minimal Residual Disease
Brief Title: Ipilimumab in Treating Patients With Relapsed or Refractory High-Risk Myelodysplastic Syndrome or Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02990; NCI-2012-02990 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NA_00076038; J1276; CDR0000744584; 9214 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); 9214 (Other: CTEP); P30CA006973 (NIH); U01CA070095 (NIH); UM1CA186691 (NIH); UM1CA186704 (NIH)
Record Dates: First submitted 2012-12-21; First posted 2012-12-31 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2017-11

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome; Previously Treated Myelodysplastic Syndrome; Recurrent Adult Acute Myeloid Leukemia; Secondary Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Ipilimumab; CTLA-4 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ipilimumab) (Experimental): INDUCTION: Patients receive ipilimumab IV on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Beginning 12 weeks after last dose of induction ipilimumab, patients receive ipilimumab IV on day 1. Treatment repeats every 12 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of ipilimumab and how well it works in treating patients with high-risk myelodysplastic syndrome or acute myeloid leukemia that has come back or no longer responds to treatment. Monoclonal antibodies, such as ipilimumab, may interfere with the ability of cancer cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and toxicity associated with the administration of ipilimumab in terms of dose limiting toxicities (DLT), and maximally-tolerated dose (MTD) in a cohort of patients with high risk myelodysplastic syndrome who failed hypomethylating therapy, and patients with acute myeloid leukemia (AML) who underwent induction therapy but are not planned for further intensive chemotherapy. (Dose-escalation) II. Determine the optimal dose of ipilimumab for the dose-expansion phase of the trial. (Dose-escalation) III. Better define immunologic profiles associated with ipilimumab use in terms of regulatory T-cells (T-regs) dynamic changes in 2 separate cohorts of myelodysplastic syndrome (MDS) and AML patients at the optimal dose level. (Dose-expansion) IV. Obtain preliminary efficacy data of ipilimumab in terms of complete response (CR), partial response (PR), and hematological improvement (HI) in both cohorts. (Dose-expansion)

SECONDARY OBJECTIVES:

I. Define immunologic profiles associated with ipilimumab use in terms of T-regs dynamic changes at different dose levels. (Dose-escalation) II. Define toxicity profiles of ipilimumab at the optimal dose in both patient cohorts. (Dose-expansion) III. Obtain preliminary data on potential correlations between noted ipilimumab-induced immunologic changes and observed toxicity and clinical responses. (Dose-expansion)

OUTLINE: This is a dose-escalation study.

INDUCTION: Patients receive ipilimumab intravenously (IV) on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Beginning 12 weeks after last dose of induction ipilimumab, patients receive ipilimumab IV on day 1. Treatment repeats every 12 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at least monthly for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Life expectancy of greater than 6 months
* Must have one of the following diagnoses:

  * Pathologically confirmed chronic myelomonocytic leukemia (CMML) or myelodysplastic syndromes (MDS) with high risk features at the time of referral for trial as defined by:

    * Intermediate (INT)-2 or high International Prognostic Scoring System (IPSS) score
    * Secondary MDS (defined as MDS developing in a patient with an antecedent hematologic disorder or any patient with prior chemotherapy or radiation exposure)
    * INT-1 MDS with excess blasts (>= 5% blasts in bone marrow [BM]) or red blood cell (RBC) transfusion-dependency
    * MDS progressing to oligoblastic acute myeloid leukemia (AML) with 21-30% BM blasts
    * CMML with >= 5% marrow blasts, or RBC or platelet transfusion-dependency, abnormal karyotype, or proliferative features (white blood cell count >=13,000/uL, splenomegaly on physical examination, or extramedullary disease)
    * All patients are required to have failed to respond or relapsed after an initial response to hypomethylating agents 5-azacitidine or decitabine or have refused to receive hypomethylating therapy; failure to respond is defined as failing to achieve a CR, PR or HI after at least 4 cycles of hypomethylating therapy; these patients could have received other therapies or not, but must have received hypomethylating therapy or have refused to receive hypomethylating therapy
  * Pathologically confirmed AML patients who have received one or two courses of induction chemotherapy or hypomethylating agent therapy AND no plans for further chemotherapy therapy, but remain with residual disease of < 5% blasts in BM, by morphology, cytogenetics, fluorescent in situ hybridization (FISH), polymerase chain reaction (PCR) or flow cytometry
* Patients must not have received any other treatment for their disease, including hematopoietic growth factors, within three weeks of beginning the trial, and should have recovered from all toxicities of prior therapy (to grade 0 or 1)
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2 at study entry ECOG, or Karnofsky >= 60%
* Calculated creatinine clearance by Modification of Diet in Renal Disease (MDRD) (CrCL) > 50 ml/min/1.73 squared meter
* Total bilirubin =< 2.0 mg/dL unless due to Gilbert's syndrome, hemolysis, or ineffective hematopoiesis
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x upper limit of normal (ULN)
* Females of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to start of ipilimumab
* Patients must have no clinical evidence of central nervous system (CNS) or pulmonary leukostasis, disseminated intravascular coagulation, or CNS leukemia
* Patients must have no serious or uncontrolled medical conditions

Exclusion Criteria:

* Any serious medical condition, uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, laboratory abnormality, or psychiatric illness/social situations that would limit compliance with study requirements or prevent the subject from signing the informed consent form
* Pregnant or breast feeding females (lactating females must agree not to breast feed while taking ipilimumab)
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Use of any other experimental drug or therapy within 21 days of baseline
* Known hypersensitivity to ipilimumab or history of allergic reactions attributed to compounds of similar chemical or biologic composition to ipilimumab
* Prior use of ipilimumab, other cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) blocking therapies, anti-programmed cell death 1 (PD 1) antibody, cluster of differentiation (CD) 137 agonist or other immune activating therapy such as anti-CD 40 antibody within the last 3 months of enrollment in the study; if any of these of these agents were used more than 3 months earlier to enrollment in study, the patient should have recovered from all toxicity and at least 3 months had passed since last use to allow for clearance and observation of any other side effects from the previous therapy
* Concurrent use of other anti-cancer agents or treatments, including other investigational agents
* Autoimmune disease: patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis]); CNS or motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre syndrome and Myasthenia Gravis, multiple sclerosis)
* Patients with known immune impairment who may be unable to respond to anti-CTLA-4 antibody
* Patients with known evidence of active cancers, or other cancer under active treatment; exceptions include patients with no evidence of disease receiving adjuvant hormone-based therapy or either breast or prostate cancer
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients with chronic human immunodeficiency virus (HIV), hepatitis B or hepatitis C infections should be excluded because of potential effects on immune function and/ or possible drug interactions
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with ipilimumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-12-14 (Actual); Primary Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of DLT of ipilimumab by grading and tabulation using National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | 42 days
Changes in percentages of T-regs | Baseline to up to 6 months post-treatment
  Changes in T-regs percentages at designated time points will be correlated with clinical responses and toxicity after ipilimumab. The response will be modeled as the vector for each individual from multiple measures of T-regs percentages as a function of time and group (MDS vs AML). T-regs percentages will be transformed onto the log-scale, and t tests will be used to compare groups at specific time points. Regression models that use generalized estimating equations will be implemented when all time points are considered to account for within-subject correlation of repeated measures.

SECONDARY OUTCOMES:
Efficacy as defined by the International working group 2006 criteria for CR, PR, HI | Up to 6 months post-treatment
  The agreement between immunologic and clinical response will be evaluated with McNemar's test, separately by cohort. Rates of CR, PR, and HI will be summarized separately by cohort and reported with an exact 95% confidence interval.
Progression free survival (PFS) | From start of study to progression or death, assessed up to 6 months post-treatment
  Median PFS will also be reported with a 95% confidence interval. As an exploratory analysis, survival endpoints will be descriptively compared with a log-rank test between patients who do and do not have an immunologic response, separately by cohort.
Overall survival (OS) | From start of study to death, assessed up to 6 months post-treatment
  Median OS will also be reported with a 95% confidence interval. As an exploratory analysis, survival endpoints will be descriptively compared with a log-rank test between patients who do and do not have an immunologic response, separately by cohort.
Rate of prior use of demethylating agents | Up to 6 months post-treatment
  Will be descriptively compared between patients who have a clinical response and by toxicity with Fisher's exact tests.
Rate of pre-treatment CR | Up to 6 months post-treatment
  Will be descriptively compared between patients who have a clinical response and by toxicity with Fisher's exact tests.
Lymphocyte counts | Baseline
  Will be summarized and compared between response and toxicity groups with either t tests or Wilcoxon rank sum tests.
T cell receptor diversity | Baseline
  Will be summarized and compared between response and toxicity groups with either t tests or Wilcoxon rank sum tests.

CONTACTS AND LOCATIONS:
Overall Officials: B. Smith, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (9):
- United States (9):
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Baylor University Medical Center, Dallas, Texas
  - Texas Oncology at Baylor Irving Cancer Center, Irving, Texas